CLINICAL TRIAL: NCT02801565
Title: Clinical Observation of Recombinant Human Growth Hormone Injection Assisted in Vitro Fertilization and Embryo Transfer (IVF-ET) in the Treatment of Polycystic Ovary Syndrome (PCOS)
Brief Title: Clinical Observation of Recombinant Human Growth Hormone Injection Assisted IVF-ET in the Treatment of PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci GH AQ CT-PCOS
Record Dates: First submitted 2016-06-06; First posted 2016-06-16 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-06

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GH AQ (Experimental): Controlled ovarian stimulation in the middle of the corpus (D21 days) of the previous menstrual cycle to use recombinant Human Growth Hormone Injection（rhGH） Injection 15IU/5mg/3mL/cartridge, 5IU per day, Subcutaneous injection after 20:00 until the HCG trigger day.
  Interventions: Drug: Conventional controlled ovarian stimulation proctol

INTERVENTIONS:
Drug: Conventional controlled ovarian stimulation proctol — Conventional controlled ovarian stimulation proctol without rhGH.

SUMMARY:
Observe validity of Recombinant Human Growth Hormone Injection assisted in IVF-ET (in vitro fertilization and embryo transfer) treatment of PCOS (polycystic ovary syndrome) patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 35 years old, married female and infertile.
* BMI≥25kg/m2.
* Diagnosed as PCOS.
* No obvious chronic organic diseases, such as liver, kidney, heart, lung, thyroid, adrenal disease.
* Subjects do not take part in other clinical trial study within 3 months.
* The subjects sign the informed consent form.

Exclusion Criteria:

* BMI<25kg/m2.
* Hyperprolactinemia and congenital adrenal cortical hyperplasia.
* Diabetes, thyroid function hyperthyroidism, thyroid dysfunction, cushing's syndrome.
* Pelvic and peritoneal tumor and tumor secreting hyperandrogenism.
* Severe acute and chronic liver and kidney disease, such as liver cirrhosis, acute and chronic renal failure, hepatitis B virus activity.
* Liver and kidney dysfunction, AST/ALT is 2.5 times higher than the normal limit, the serum of creatinine is 2 times higher than the normal level.
* Diseases affecting outcome of IVF pregnancy, eg, hydrosalpinx, hysteromyoma>4 cm, adenomyosis, endometriosis, endometrial cyst of ovary, unilateral ovary, tuberculosis of reproductive system.
* Allergic to E. coli. expression product and its excipients.
* Being involved in other drug clinical researchers.
* The researchers consider who is not suitable for the group.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | One year
Number of fertilized oocytes | One year

SECONDARY OUTCOMES:
Number of retrieved oocytes | One year
Number of high quality embryos | One year
Number of transferred embryos | One year

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China